CLINICAL TRIAL: NCT05592561
Title: Impact of Caffeine, Theanine, Tyrosine Ingestion on Markers of Stress in Response to a Cognitive Challenge and Virtual Reality Active Shooter Drill
Brief Title: Impact of Supplements on Stress Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Collaborators: M. Hunter Martaindale (Unknown); C. Dillard (Unknown); D. Gonzalez (Unknown)
Responsible Party: Principal Investigator, Matt McAllister, Associate Professor, Texas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Supplements and VR-ASD
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Physiological Stress

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of four treatments:
  1. placebo ingestion
  2. caffeine ingestion
  3. theanine ingestion
  4. tyrosine ingestion
  nutrient ingestion takes place 40 min prior to being exposed to a mental stress task.
Who Masked: Participant
Masking Description: The researchers will prepare the caffeine, placebo, tyrosine, and theanine containing sweetened and flavor matched beverages immediately before subjects ingested them. The subjects will not be told which treatment they will be receiving. There will be no indicative labels on the water bottle provided to them which contained the crystal light which will be mixed with either 200 mg of caffeine, 200 mg of theanine, 2000 mg tyrosine or crystal light only (placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caffeine group (Experimental): Subjects will receive 200 mg of caffeine powder which was obtained from a 200 mg capsule (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada). Researchers will break open the capsule and mix with water and 5/8 tsp of crystal light immediately before subjects ingest the randomly assigned treatment.
  Interventions: Other: mental stress task
- Placebo (Placebo Comparator): flavored water (sweetened with crystal light powder, 0.5 tsp) will be provided to subjects without any caffeine powder added.
  Interventions: Other: mental stress task
- Theanine group (Experimental): 200mg pure theanine powder (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada) + 8 oz water+ 0.55 tsp crystal light will be ingested.
  Interventions: Other: mental stress task
- Tyrosine group (Experimental): 2000 mg pure tyrosine powder (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada) +8 oz water + 0.5 tsp crystal light will be ingested.
  Interventions: Other: mental stress task

INTERVENTIONS:
Other: mental stress task — The stress protocol used for this experiment utilized a cognitive challenge and a previously studied virtual reality active shooter drill (VR-ASD). The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). Immediately upon completion of the cognitive challenge, the subjects completed the VR-ASD scenario (~2 min) followed by the same cognitive challenge with different questions (another 4 min). The total duration was ~10 min.

SUMMARY:
The goal of this clinical trial is to examine the effects of caffeine, theanine and tyrosine ingestion on markers of stress in healthy college aged individuals that are exposed to a mental stress task. The main questions to answer are:

1. what is the impact of a mental stress task involving a cognitive challenge and virtual reality based active shooter scenario on markers of subjective and biological stress?
2. what is the impact of supplement ingestion (caffeine, theanine, tyrosine, analyzed separately) 40 min prior to exposure to the mental stress task?

DETAILED DESCRIPTION:
This study will take place in two blocks of randomization, where during the first segment of randomization, participants will be randomly assigned to ingest either 200mg of caffeine powder or a placebo beverage (0mg caffeine) which will be flavored and sweetened with crystal light powder. Ingestion takes place 40 min prior to engaging in a mental stress task which included a cognitive challenge and a virtual reality based active shooter drill. Researchers will compare the two treatment groups in terms of changes in heart rate, subjective stress, and salivary markers of stress before and after the mental stress task.

During the second block of randomization, subjects will be randomly assigned to ingest either 200 mg of theanine powder or 2000 mg of tyrosine powder with crystal light powder, mixed with water, also 40 min prior to the same mental stress task. The placebo condition from the first block of randomization will be used as a control for comparison for all three supplements. The experimental procedures are the same for all four treatments (placebo, caffeine, tyrosine, theanine) and only differ with respect to which beverage was ingested prior to the mental stress task.

All procedures were reviewed and approved by the University Institutional Review Board.

Experimental Procedures Upon arrival to the testing site, body mass will be measured using a digital scale (Rice Lake Weighing Systems, Rice Lake, WI, USA), and height will be measured using a portable stadiometer (213; SECA, CA, USA). Subjects will be then instructed to rinse their mouth with water and rest in a quiet room for 10 minutes. During this time, they will be equipped with a heart rate (HR) monitor (Polar verity sense; Polar Electro Ltd, Kempele, Finland). Immediately after the 10 minute rest period, an initial saliva sample, HR and SAI measures were collected (45 min prior to mental stress task). Five min after this (40 min pre mental stress task), subjects will consume their assigned treatment: either the placebo (crystal light + 8 oz of water) or caffeine supplement (200 mg caffeine + crystal light + 8 oz of water ). Throughout the experimental session, HR, SAI, and saliva samples will be collected a total of four times: 1) 45 minutes prior to the start of the mental stress task, 2) immediately before the mental stress task, 3) immediately after the mental stress task, and 4) 30 min after the mental stress task.

Mental Stress Task: Cognitive Challenge & VR-ASD The stress protocol used for this experiment will utilize a cognitive challenge and a previously studied VR-ASD. The cognitive challenge will include a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). Immediately upon completion of the cognitive challenge, the subjects will complete the VR-ASD scenario (~2 min) followed by the same cognitive challenge with different questions (another 4 min). The total duration was ~10 min.

Stroop Challenge For the Stroop challenge, the subjects will be presented with a 0.5 second display of a word on the computer screen (i.e., yellow, green, red, or blue). However, the word is written in conflicting-color font presenting a mental conflict. Subjects are required to identify the text font color as quickly as possible using a color-coded keypad. Note, 0.5 seconds was allowed for the response. Feedback included total attempts, total correct and incorrect responses, missed responses, and response time.

Arithmetic Calculations The arithmetic calculations consisted of addition and subtraction with single, double-, and triple-digit numbers (e.g., 736 minus 58). The subject was given 10 seconds to respond to each mathematical question. Failure to respond within the allotted time resulted in an incorrect response. The subjects were presented with 2-min of the Stroop Challenge followed by 2-min of mental arithmetic. This will occur both before and after the VR-ASD.

Virtual Reality Active Shooter Drill The general procedures for the VR-ASD are previously described and based on a live -action ASD protocol (McAllister et. al., 2020). Briefly, the subject advanced down a ~3-meter-long hallway where two wounded victims were encountered. A white female victim with traumatic injuries was laying on the ground while an African American female victim "ran" out of a classroom with a gunshot wound to the left arm and leg. Upon arriving to the classroom, the subject observed a white female on the ground with a traumatic head injury as well as the shooter (white male) firing a handgun at an African American male. The subject was required to fire his/her weapon to prevent the shooter from turning toward the subject and eliciting a response. Once the shooter fell down after being shot by the subject, the VR-ASD scenario ended. The VR-ASD was presented using HTC VIVE Pro VR equipment (HTC Corp, New Taipei, Taiwan). The VR laboratory environment is larger than the virtual environment (~35 ft x 20 ft); therefore, subjects are able to physical maneuver throughout the ASD without disruption.

Supplement Ingestion Caffeine supplement capsules containing 200 mg caffeine powder (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada)will be used for the present study. The capsules will be broken into halves and the caffeine powder inside was mixed with 8 oz of water and calorie free crystal light. For the placebo treatment, the same flavor of crystal light will be mixed with 8 oz of water.add that the treatments were flavor/sweetness matched.

For the theanine treatment, 200mg pure theanine powder (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada) will be mixed with 8 oz water and crystal light

for the tyrosine treatment, 2000mg of tyrosine powder (Hard Eight Nutrition, LLC, dba, Bulk Supplements, Henderson, Nevada) will be mixed with 8oz of water and crystal light.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy, aged 18-40,
* free from any known cardiovascular or metabolic diseases,
* free from any major stressors within the last 30 days such as birth of a child, abortion, or divorce.

Exclusion Criteria:

* subjects are required to not have a history of motion sickness or vertigo,
* not previously diagnosed with a brain injury or epilepsy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
salivary secretory IgA | Up to 10 months
  SIgA is a marker of immune function and salivary SIgA concentrations tend to increase when exposed to stress
salivary alpha amylase | Up to 10 months
  salivary alpha amylase is an enzyme involved in digestive processes. amylase concentrations in saliva have been shown to reflect sympathetic stress. Thus, as sympathetic stress increases, salivary alpha amylase concentrations tend to increase
salivary cortisol | Up to 10 months
  salivary cortisol is a marker of stress which reflects activation of the hypothalamic pituitary adrenal axis.
heart rate | Up to 10 months
  heart rate reflects activity from the parasympathetic and sympathetic nervous system and increases when exposed to stress
State anxiety inventory | Up to 10 months
  state anxiety inventory is a subjective scale which includes six short statements such as "I feel calm" or " I feel tense" and composite scores of participant responses are used for analysis. Higher values reflect higher subjective anxiety.

SECONDARY OUTCOMES:
mental arithmetic incorrect | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.
mental arithmetic missed responses | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.
mental arithmetic response time | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.
Stroop challenge number of incorrect | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.
Stroop challenge number of missed responses | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.
Stroop challenge response time | Up to 10 months
  The cognitive challenge included a modified version of the Stroop challenge (2 min) and mental arithmetic calculations (2 min) presented to the subject via e-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA, USA). The software included number of correct, incorrect, missed responses and response time.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State University, San Marcos, Texas, United States

REFERENCES:
- [Derived] McAllister MJ, Martaindale MH, Dillard CC, McCullough R. Impact of L-theanine and L-tyrosine on markers of stress and cognitive performance in response to a virtual reality based active shooter training drill. Stress. 2024 Jan;27(1):2375588. doi: 10.1080/10253890.2024.2375588. Epub 2024 Jul 8. PMID 38975711
- [Derived] McAllister MJ, Martaindale MH, Dillard CC, Gonzalez DE. Stress response to virtual reality based active shooter training: Impact of caffeine consumption. Psychoneuroendocrinology. 2024 Mar;161:106923. doi: 10.1016/j.psyneuen.2023.106923. Epub 2023 Dec 7. PMID 38142605